CLINICAL TRIAL: NCT06911827
Title: A Phase Ib/II Open-Label, Dose-Escalation and Dose-expansion Clinical Study to Evaluate the Safety, Pharmacokinetics, Immunogenicity and Efficacy of QLP2117 in Combination With QL2107 in Advanced Solid Tumor Patients
Brief Title: A Study of QLP2117 in Combination With QL2107 in Advanced Solid Tumor Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLP2117-201
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ib/II (Experimental): * Experimental: Ib： QLP2117 in combination with QL2107 Dose escalation and PK expansion
  * Experimental: II： QLP2117 in combination with QL2107 Dose expansion
  Interventions: Drug: QLP2117; Drug: QL2107

INTERVENTIONS:
Drug: QLP2117 — Specified dose on specified days
Drug: QL2107 — Specified dose on specified days

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of QLP2117 in combination with QL2107 in Advanced Solid Tumor Patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of recurrent or refractory advanced solid tumours, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
* At least one measurable disease for expansion cohorts per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1(phase Iba dose escalation only requires at least one assessable lesion)
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Agree to provide archived tumor tissue samples of primary or metastatic lesions.
* Have adequate organ function as described in the protocol.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* HBsAg/HBcAb positive and HBV-DNA>1000 copy/mL;HCV-Ab positive and detection of HCV-RNA suggested viral replication
* Is currently participating and receiving study medication in another study within 4 week prior to the first dose of study treatment
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has an active infection requiring systemic therapy
* Has received a live vaccine wihtin 30 days of planned start of study treatment
* Known history of, or any evidence of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 21days
Percentage of Participants Experiencing Adverse Events (AEs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | up to 96 weeks
Objective Response Rate for phase II | up to 96 weeks